CLINICAL TRIAL: NCT01731678
Title: Transcranial Magnetic Stimulation for Adolescent Depression
Acronym: TMSAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Frank MacMaster, PhD, Cuthbertson and Fischer Chair in Paediatric Mental Health, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-24656
Record Dates: First submitted 2012-11-03; First posted 2012-11-22 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Masking Description: Open label rTMS
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial Magnetic Stimulation (Experimental): The standardized treatment location will be the left DLPFC. Anatomical T1 images from the pre-intervention MRI will be loaded into our Transcranial Magnetic Stimulation (TMS) lab neuronavigation software (Brainsight2, Rogue Research, Montreal). Following 3D co-registration of the TMS coil with the patient's MRI images and head, the coil will be placed over the left DLPFC (tangential to scalp, angle of 45 degrees to midline). Interventional repetitive TMS (rTMS) (Magstim Rapid2, Wales, UK) will consist of 40 suprathreshold (120% RMT) pulses over 4 seconds (10 Hz) with an inter-train interval of 26 seconds. Treatment sessions will last 37.5 minutes (75 trains/3000 pulses). Treatments will occur on each weekday for three weeks (15 days total).
  Interventions: Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — The standardized treatment location will be the left DLPFC. Anatomical T1 images from the pre-intervention MRI will be loaded into our Transcranial Magnetic Stimulation (TMS) lab neuronavigation software (Brainsight2, Rogue Research, Montreal). Following 3D co-registration of the TMS coil with the patient's MRI images and head, the coil will be placed over the left DLPFC (tangential to scalp, angle of 45 degrees to midline). Interventional repetitive TMS (rTMS) (Magstim Rapid2, Wales, UK) will consist of 40 suprathreshold (120% RMT) pulses over 4 seconds (10 Hz) with an inter-train interval of 26 seconds. Treatment sessions will last 37.5 minutes (75 trains/3000 pulses). Treatments will occur on each weekday for three weeks (15 days total).

SUMMARY:
Major depression (or MDD) in adolescents is a major public health problem. MDD affects approximately 15% of adolescents; it is associated with impairment in social, family, and academic functioning, and it is a major risk factor for suicide - a leading cause of death in adolescents . Unfortunately, there is a paucity of treatment options for this age group. Selective serotonin reuptake inhibitors (SSRIs) are the only class of medications approved for treating MDD in adolescents, but rates of remission following treatment with SSRIs are only 30 to 45 percent. Cognitive behavior therapy is associated with similar remission rates and access is limited. Most adolescents will require more than one therapeutic intervention in order to achieve full symptom control. Collectively, there is overwhelming evidence that additional treatment options are urgently needed to improve outcomes for teens with MDD. One novel treatment for adolescent MDD is repetitive transcranial magnetic stimulation (rTMS). Studies in children have been limited (a total of 23 cases). This is surprising given the evidence suggesting younger adult subjects with MDD respond better to rTMS (56% response rate) than older subjects. This limited experience with rTMS for adolescent MDD represents a substantial gap in the knowledge, recently recognized in publications calling for further study of rTMS in adolescent depression. Most importantly, the mechanism of action of rTMS in adolescent MDD is not well understood. The objective of this application is to develop an understanding of the brain alterations associated with the positive clinical changes that occur with rTMS in adolescent MDD. Such knowledge will provide the basis for pursuing rTMS for adolescent MDD as a rational therapeutic technique.

Specific Aim: To compare the effect of rTMS on DLPFC glutamate concentration in adolescent MDD. The investigators hypothesize an increase (normalization to controls) in DLPFC glutamate after three weeks of rTMS. Furthermore, the change in glutamate concentration will correlate with a change in MDD symptoms.

DETAILED DESCRIPTION:
PURPOSE: The purpose of this study is to identify neuroimaging, physiological, and clinical predictors of response, remission, and recovery to repetitive transcranial magnetic stimulation in youth with treatment resistant major depressive disorder.

BACKGROUND: Major depressive disorder (MDD) is a major public health problem in adolescents. Unfortunately, there are no effectively targeted treatment options for this age group. Current remedies are limited in their effectiveness in youth with response and remission rates no greater than 60 to 30% respectively and treatment effects are not sustained throughout the life cycle. Further, ongoing controversies persist regarding the safety of antidepressants in youth. Current interventions were developed to solely target the symptoms of rather than the underlying neurobiology. Most importantly, there is no way to accurately predict an individual patient's response to interventions. Consequently, there is a critical need for optimally targeted interventions that directly address the relevant pathophysiology of depression.

Repetitive transcranial magnetic stimulation (rTMS) targeting the left dorsolateral prefrontal cortex (DLPFC) is effective in adults with depression. rTMS is twice as likely to result in response (relative risk or RR: 2.35 [95% confidence interval or CI: 1.70-3.25]) and remission (RR: 2.24 [95% CI: 1.53-3.27] than a sham procedure Evidence in youth is also encouraging, with a 66% response rate in our pilot data (see Summary of Progress). The DLPFC plays a critical role in emotional regulation, directly connecting it to depressive symptomology. Our lab and others have clearly implicated structural and functional deficits in the DLPFC in youth with MDD. What is not known is what biomarkers best predict response, remission, and recovery with rTMS in youth with treatment resistant MDD. As response is not universal, this is a significant gap in our knowledge. Our basic model is that rTMS increases expression of BDNF, up-regulates activity of endocannabinoids, increases glutamate concentrations, and increases DLPFC activity - correcting the deficit seen in MDD. These biologic changes enhance executive control of mood state (see our pilot data in the Summary of Progress). These positive effects may be moderated by comorbidity (i.e., social phobia) and genotype (i.e., BDNF). How this model fits with response, remission, and recovery has yet to be fully tested and this information has the potential to be directly clinically meaningful. The central aim of the project is to evaluate predictors of rTMS response, remission, and recovery based on integrated neuroimaging, physiological, and clinical measures. While not a clinical trial per se (efficacy is not the primary outcome measure), we will use a non-randomized sham lead in to a single active (rTMS) arm study design as a framework for biomarker discovery.

To accomplish this goal, we will pursue the following specific aims: The primary aim is to identify baseline neuroimaging, physiological, and clinical predictors of response to 3 weeks of rTMS treatment in adolescents with treatment resistant MDD.

ELIGIBILITY:
Inclusion Criteria:

* age (12-22 years),
* MDD failing to respond to at least one SSRI trial (minimum 8 weeks treatment at an adequate dose; determined retrospectively), and
* informed consent. Healthy controls with no psychiatric history (who do not receive rTMS) will undergo MRI scans to allow for comparison with MDD patients.

Exclusion Criteria:

* previous seizures or epilepsy,
* hypertension,
* additional neurological or psychiatric diagnoses (specifically: bipolar disorder, psychosis, pervasive developmental disorder, eating disorders, and post-traumatic stress disorder).

As 3T MRI will be used, pregnancy is exclusionary.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank P MacMaster, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] MacMaster FP, Croarkin PE, Wilkes TC, McLellan Q, Langevin LM, Jaworska N, Swansburg RM, Jasaui Y, Zewdie E, Ciechanski P, Kirton A. Repetitive Transcranial Magnetic Stimulation in Youth With Treatment Resistant Major Depression. Front Psychiatry. 2019 Mar 29;10:170. doi: 10.3389/fpsyt.2019.00170. eCollection 2019. PMID 30984044

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Magnetic Stimulation: The standardized treatment location is the left DLPFC. Anatomical T1 images from the pre-intervention MRI were loaded into our neuronavigation software (Brainsight2, Rogue Research, Montreal). The coil was placed over the left DLPFC (tangential to scalp, angle of 45 degrees to midline). Interventional repetitive TMS (rTMS) (Magstim Rapid2, Wales, UK) consisted of 40 suprathreshold (120% RMT) pulses over 4 seconds (10 Hz) with an inter-train interval of 26 seconds. Treatment sessions will last 37.5 minutes (75 trains/3000 pulses). Treatments will occur on each weekday for three weeks (15 days total).
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation
Started | 39
Completed | 32
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Did not meet inclusion criteria | 1
Not completed — RMT too high, making TMS difficult | 3

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17.57 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 32
Baseline Hamilton Depression Rating Scale Score [Mean (Standard Deviation); unit: units on a scale] — Name: Hamilton Depression Rating Scale Construct: Depression Range: 0-52 Direction: Higher is worse depression symptoms/severity Sub-scales: Not applicable. Reference: Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96.
  units on a scale | 20.25 (6.37)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale
Description: Response defined as: a reduction of Hamilton Depression Rating Scale score of 50% or more Name: Hamilton Depression Rating Scale Construct: Depression Range: 0-52 Direction: Higher is worse depression symptoms/severity Sub-scales: Not applicable. Reference: Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96.
Time Frame: Three weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 32
score on a scale | 9.38 (5.44)

2. Other Pre Specified Outcome: Interim Analysis - rTMS Tolerability Scale
Description: There will be an interim analysis to review safety, tolerability (as measured by our rTMS tolerability scale) after the first 10 rTMS patients. Should there be significant concerns, the team will terminate the study. Ten was selected as it is close to previous reports and should be informative.
Time Frame: After the first 10 patients are completed
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Interim Analysis - Ham-D
Description: There will be an interim analysis to review response (Ham-D) after the first 10 rTMS patients. Should there be significant concerns, the team will terminate the study. Ten was selected as it is close to previous reports and should be informative.
Time Frame: After the first 10 patients are completed
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Six weeks
Description: We used a TMS tolerability scale to monitor participants weekly.
Arm/Group | Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2012-04-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT01731678/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2012-04-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT01731678/Prot_SAP_001.pdf